CLINICAL TRIAL: NCT04019145
Title: Clinical Evaluation of Fiber Reinforced Bulk Fill Resin Composite Versus Incremental Packing of Nanohybrid Resin Composite in Restoration of Deep Proximal Lesions of Permanent Posterior Molars: A Randomized Controlled Trial
Brief Title: Clinical Evaluation of Fiber Reinforced Resin Composite Base Versus Incremental Packing of Nanohybrid Resin Composite
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Salem, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28909092104862
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Caries Class II
MeSH Terms: interventions — EverX Posterior; Composite Resins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Reinforced bulk fill resin composite (Experimental): Fiber reinforced bulk fill resin composite dentine substitute, capped occlusally and proximally (closed centripetal technique) by nanohybrid resin composite.
  Interventions: Drug: EverX Posterior
- nanohybrid resin composite incrementation (Active Comparator): Nanohybrid resin composite layering to fill the whole cavity, using closed centripetal technique.
  Interventions: Drug: Resins, Composite

INTERVENTIONS:
Drug: EverX Posterior — fiber reinforced bulk fill resin composite
  Other Names: Fiber reinforced bulk fill dentine substitute
  Arms: Fiber Reinforced bulk fill resin composite
Drug: Resins, Composite — incremental packing of Nanohybrid Resin composite
  Other Names: Universal Restorative Nanohybrid resin composite
  Arms: nanohybrid resin composite incrementation

SUMMARY:
A clinical trial, comparing two different incrementation techniques in the restoration of proximal caries in permanent posterior teeth . One utilizes a fiber reinforced bulk fill base material, followed by an occlusal nanohybrid capping layer. The other utilizes incremental packing of nanohybrid resin composite material to fill the whole cavity.

DETAILED DESCRIPTION:
The aim of this study is to conduct an RCT to evaluate the clinical performance of the fiber reinforced bulk fill resin composite in comparison to incremental packing of nanohybrid resin composite.

Examination and selection of all patients will be done according to inclusion and exclusion criteria. Diagnosis of patients' chief complaint and teeth that will be involved in this study will be done. Teeth are to be chosen according to standardized radiographic examination. Teeth should have proximal, primary deep carious lesions involving 2/3 of the entire dentin thickness with no continuity between the carious cavity and the pulp chamber.

A Class II cavity will be prepared after local anesthesia has been given as required. The cavity will be prepared using a high-speed hand-piece with air and water coolant and diamond burs of different sizes. Sharp excavators will allow accessible removal of soft carious lesions will be used. Any tooth that will suffer from pulpal exposure will be excluded from the study. Finishing of the cavity walls will be done using a fine-grit, yellow coded, diamond bur.

Rubber dam isolation will be done.

Sectional matricing and wedging will be done. Followed by, placement of restorative material according to the randomization sequence.

A closed centripetal technique will be utilized, where a proximal wall will be built using nanohyrbid resin composite first, followed by filling of cavity with bulk-fill fiber reinforced resin composite material in increments of 3-4mm, as required to end up with leaving an occlusal space on top of at least 2mm. Then, an occlusal increment of nanohybrid resin composite will be applied. Finally finishing and occlusal adjustment will be done under water spray by using superfine diamond burs. Polishing will be done using pre-impregnated rubber cups. Materials will be manipulated according to manufacturer instructions.

A closed centripetal, oblique incrementation technique will be used to completely fill the whole cavity. Increments should be of 2mm thickness or less and should be placed obliquely from the cavity walls. Then finishing and occlusal adjustment will be done under water spray by using superfine diamond burs. Polishing will be done using pre-impregnated rubber cups. Materials will be manipulated according to manufacturer instructions

Outcome Measuring Device: modified USPHS criteria .

Primary Outcomes:

Mechanical evaluation:

Fracture and Retention Marginal integrity Marginal Discoloration Anatomic Form Surface Texture Proximal Contact Radiographic Examination

Secondary Outcomes:

Biological evaluation:

Postoperative Sensitivity Recurrent Caries

ELIGIBILITY:
Inclusion Criteria:

Patient-related criteria:

* Patients consulting in one of the outpatient clinic listed above.
* Able to tolerate necessary restorative procedures.
* Provide informed consent.
* Accepts the one year follow-up period.

Tooth related criteria:

* Teeth with primary deep carious lesions involving 2/3 of the entire dentin thickness with no continuity between the carious cavity and the pulp chamber.
* Teeth are vital according to pulp-sensitivity tests.

Exclusion Criteria:

Patient-related criteria:

* Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.
* Pregnant women; as radiographs cannot be taken for them.
* Allergy to any of the restorative materials, including anesthetics.
* Uncooperative patients, will not abide by the instructions or attend the appointments.

Tooth related criteria:

* Deciduous teeth; as the study is targeting only permanent teeth.
* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests), which would indicate irreversible pulpal damage.
* Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion, which would indicate pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Mechanical outcome according to USPHS criteria | 12 months
  fracture or retention, marginal integrity, marginal discoloration, anatomic form, proximal contact, radiographic examination and surface texture

SECONDARY OUTCOMES:
Biological outcome according to USPHS criteria | 12 months
  postoperative sensitivity and recurrent caries

CONTACTS AND LOCATIONS:
Overall Officials: Olfat Hassanein, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No